CLINICAL TRIAL: NCT03822871
Title: A Phase 1 Trial for Evaluation of Safety and 177Lu Radiation Dosimetry of CTT1403: A Peptidomimetic Inhibitor of Prostate Specific Membrane Antigen, in Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: A Trial of CTT1403 for Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Targeted Technology (Industry)
Collaborators: University of California, San Francisco (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTT1403-101; 5R44CA239461-06 (NIH)
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; metastatic castration resistant prostate cancer; prostate specific membrane antigen; mCRPC; PSMA; positron emission tomography; PET; radiotherapy; targeted therapy; lutetium; 177Lu
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Escalating doses of 0.75 GBq - 2.0 GBq of CTT1403
  Interventions: Drug: CTT1403; Drug: CTT1057; Drug: 68Ga-PSMA-11
- Dose Escalation/Expansion (Experimental): Escalating doses of 3.0 GBq - 9.0 GBq of CTT1403
  Interventions: Drug: CTT1403; Drug: CTT1057; Drug: 68Ga-PSMA-11

INTERVENTIONS:
Drug: CTT1403 — Escalating doses of 0.75 GBq - 9.0 GBq will be administered in an accelerated to traditional 3+3 dose escalation design. After escalation, 10 additional patients will be enrolled into a dose expansion cohort. Patients meeting eligibility criteria with demonstrated cessation of disease progression will be offered a second dose of the study drug, CTT1403.
Drug: CTT1057 — Patients will be screened with CTT1057 or 68Ga-PSMA-11 PSMA PET to demonstrate presence of at least 3 PSMA avid lesions that can be targeted by the study drug, CTT1403. 5-7 weeks after administration of study drug, patients will be evaluated a second time with PSMA PET imaging using with either CTT1057 or 68Ga-PSMA-11 to assess potential efficacy of CTT1403.
Drug: 68Ga-PSMA-11 — Patients will be screened with CTT1057 or 68Ga-PSMA-11 PSMA PET to demonstrate presence of at least 3 PSMA avid lesions that can be targeted by the study drug, CTT1403. 5-7 weeks after administration of study drug, patients will be evaluated a second time with PSMA PET imaging using with either CTT1057 or 68Ga-PSMA-11 to assess potential efficacy of CTT1403.

SUMMARY:
The purpose of this study is to find the highest dose level of study drug, CTT1403, that can be safely administered to patients with metastatic castration resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This is a Phase 1, first-in-human dose escalation/dose expansion study evaluating escalating doses of CTT1403 in patients with PSMA-avid mCRPC with progressive disease on at least one androgen signaling inhibitor, followed by a dose expansion to further evaluate the safety, tolerability, efficacy and biological activity of CTT1403. CTT1403 is a PSMA-targeted 177Lu-labeled radiotherapy being developed for prostate cancer with a unique PSMA binding scaffold and an albumin binding moiety to extend circulation half-life. The PSMA binding scaffold is shared with CTT1057, a PSMA-specific PET diagnostic imaging agent shown in Phase 1 clinical trials to be specifically taken up by PSMA+ tumor. PSMA PET imaging by CTT1057 will be used diagnostically to select patients with PSMA-avid disease for treatment. The purpose of this study is to identify the dose limiting toxicity and recommended phase 2 dose of CTT1403. Eligible participants with demonstrated therapeutic benefit will be offered a second dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed prostate adenocarcinoma that is metastatic and castration resistant (mCRPC).
* At least 3 metastatic foci avid for PSMA-specific PET agent (CTT1057) uptake on Screening PSMA PET.
* Has received docetaxol, ineligible for docetaxol, or refused docetaxol for the treatment of prostate cancer.
* Has progression by the PCWG3 criteria during or after treatment with either abiraterone or enzalutamide
* Male Age ≥ 18 years.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (see Appendix 2).
* Demonstrate adequate organ function

Exclusion Criteria:

* Has received previous treatment with radium-223 or another radiopharmaceutical within 3 months prior to first dose of CTT1403.
* Has received prior systemic anti-cancer therapy (excluding radiopharmaceutical) within 14 days, or 5 half-lives, whichever is shorter, prior to first dose of CTT1403.
* Has received external-beam radiation within 14 days prior to first dose of CTT1403.
* Has received cabazitaxel for the treatment of mCRPC.
* Has received previous treatment with a therapeutic targeting PSMA.
* Has an additional active malignancy requiring therapy that may confound the assessment of the study endpoints.
* Has clinically significant cardiovascular disease
* Has a history of untreated brain metastases
* Has evidence of diffuse bone marrow involvement by prostate cancer in the judgment of study investigator.
* Clinically significant urinary obstruction or moderate/severe hydronephrosis on baseline imaging.
* Has a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days before CTT1403 administration.
* Has known positive status for chronic hepatitis B or hepatitis C
* Known or suspected myelodysplastic syndrome.
* Has any medical condition which in the opinion of the Investigator places the patient at an unacceptably high risk for toxicities.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer is a disease only occurring in males.
Enrollment: 17 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2023-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Langton-Webster, PhD, Study Chair — Cancer Targeted Technology; Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.75 GBq Cohort: 0.75 GBq dose of CTT1403
- 1.5 GBq Cohort: 1.5 GBq dose of CTT1403
- 2.0 GBq Cohort: 2.0 GBq dose of CTT1403
- 3.0 GBq Cohort: 3.0 GBq dose of CTT1403
- 4.5 GBq Cohort: 4.5 GBq dose of CTT1403
- 6.0 GBq Cohort: 6.0 GBq dose of CTT1403
- 7.5 GBq Cohort: 7.5 GBq dose of CTT1403
- 9.0 GBq Cohort: 9.0 GBq dose of CTT1403
Period: Overall Study
Arm/Group | 0.75 GBq Cohort | 1.5 GBq Cohort | 2.0 GBq Cohort | 3.0 GBq Cohort | 4.5 GBq Cohort | 6.0 GBq Cohort | 7.5 GBq Cohort | 9.0 GBq Cohort
Started | 1 | 1 | 1 | 3 | 4 | 3 | 3 | 1
Completed | 1 | 1 | 1 | 3 | 4 | 3 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2.0 GBq Cohort: 2.0GBq dose of CTT1403
- Total: Total of all reporting groups
Arm/Group | 0.75 GBq Cohort | 1.5 GBq Cohort | 2.0 GBq Cohort | 3.0 GBq Cohort | 4.5 GBq Cohort | 6.0 GBq Cohort | 7.5 GBq Cohort | 9.0 GBq Cohort | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 3 | 3 | 1 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 83 | 75 | 79 | 65 (7.55) | 70 (2.58) | 72 (7.81) | 82 (1.00) | 74 | 73.41 (7.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 1 | 1 | 1 | 3 | 4 | 3 | 3 | 1 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 1 | 1 | 3 | 3 | 3 | 3 | 1 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 0 | 3 | 3 | 3 | 3 | 1 | 15
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 3 | 4 | 3 | 3 | 1 | 17

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Dose-limiting Toxicity at Escalating Dose Levels of CTT1403
Description: The dose-limiting toxicity was defined as any of the following:
  1. Grade 4 neutropenia lasting > 5 consecutive days
  2. Grade 3 or 4 febrile neutropenia
  3. Grade 4 thrombocytopenia lasting ≥ 7 days, or Grade 3 or 4 thrombocytopenia with clinically significant bleeding or requirement for platelet transfusion
  4. Any nonhematologic, treatment-related AE ≥ Grade 3, with the exceptions of Grade 3 nausea, vomiting, diarrhea, non-clinically significant electrolyte abnormality, constipation, fever, fatigue, or skin rash that resolves to Grade ≤ 2 within 72 hours with optimal medical management
  5. Any other treatment-related toxicity that results in delay of Cycle 2 administration of CTT1403 by > 21 days and/or toxicity considered by the Investigator and Sponsor's medical representatives to be dose-limiting.
Time Frame: 6-8 weeks from time of injection on Cycle 1 - Day 1
Measure: Count of Participants; unit: Participants
Groups:
- 0.75 GBq Cohort: 0.75 GBq dose of CTT1043
- 1.5 GBq Cohort: 1.5 GBq dose of CTT1043
- 2.0 GBq Cohort: 2.0 GBq dose of CTT1043
- 3.0 GBq Cohort: 3.0 GBq dose of CTT1043
- 4.5 GBq Cohort: 4.5 GBq dose of CTT1043
- 6.0 GBq Cohort: 6.0 GBq dose of CTT1043
- 7.5 GBq Cohort: 7.5 GBq dose of CTT1043
- 9.0 GBq Cohort: 9.0 GBq dose of CTT1043
Arm/Group | 0.75 GBq Cohort | 1.5 GBq Cohort | 2.0 GBq Cohort | 3.0 GBq Cohort | 4.5 GBq Cohort | 6.0 GBq Cohort | 7.5 GBq Cohort | 9.0 GBq Cohort
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 3 | 3 | 1
Participants
  Number of participants who experienced a dose-limiting toxicity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants who did not experience a dose-limiting toxicity | 1 | 1 | 1 | 3 | 4 | 3 | 3 | 1

2. Primary Outcome: Objective Response Rate by RECIST v1.1 Criteria
Description: Changes in only the largest diameters (unidimensional measurment) of the tumor lesions are used in the RECIST v1.1 criteria. Data presented as RECIST Overall Response.
Time Frame: Cycle 1-Day 35, Cycle 2-Day 35, 30 Days After Last Dose, 8 Weeks Post-Treatment. Each cycle lasted 35 days.
Population: In cases where the number analyzed differs from the total number in the group, data was either not available, patient was lost to follow-up, or patient withdrew.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.75 GBq Cohort | 1.5 GBq Cohort | 2.0 GBq Cohort | 3.0 GBq Cohort | 4.5 GBq Cohort | 6.0 GBq Cohort | 7.5 GBq Cohort | 9.0 GBq Cohort
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 3 | 3 | 1
Participants
  Number of patients with stable disease on Cycle 1-Day 35 | 0 | 1 | 0 | 1 | 4 | 2 | 1 | 1
  Number of patients with progressive disease on Cycle 1-Day 35 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0
  Number of patients with stable disease on Cycle 2-Day 35 | 0 | 1 | 0 | 0 | 2 | 1 | 3 | 0
  Number of patients with progressive disease on Cycle 2-Day 35 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
  Number of patients with stable disease 30 days after last dose | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of patients with progressive disease 30 days after last dose | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Number of patients with stable disease 8 weeks post-treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of patients with progressive disease 8 weeks post-treatment | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0

3. Secondary Outcome: Assessment of Organ Dosimetry of CTT1403 by SPECT/CT Imaging
Description: Organ dosimetry was assessed via SPECT/CT imaging until two imaging periods have been collected in which study drug cannot be detected by SPECT/CT. Time points included (2 hrs ± 1 followed by 24±12 hrs, 48±12 hrs, and 168±24 hrs post-infusion on Cycle 1-Day 1. Data calculated using OLINDA. Absorbed dose is calculated as single value wherein absorbed dose is proportional to the integral of activity over time.
Time Frame: 2 hrs ± 1 followed by 24±12 hrs, 48±12 hrs, and 168±24 hrs post-infusion on Cycle 1-Day 1
Measure: Mean (Standard Deviation); unit: Gy/GBq
Arm/Group | 0.75 GBq Cohort | 1.5 GBq Cohort | 2.0 GBq Cohort | 3.0 GBq Cohort | 4.5 GBq Cohort | 6.0 GBq Cohort | 7.5 GBq Cohort | 9.0 GBq Cohort
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 3 | 3 | 1
Gy/GBq
  Mean absorbed dose per GBq - Left Kidney | 0.608 | 0.611 | 0.760 | 1.024 (0.428) | 0.579 (0.127) | 0.518 (0.072) | 0.774 (0.199) | 0.699
  Mean absorbed dose per GBq - Right Kidney | 0593 | 0.585 | 1.021 | 1.032 (0.550) | 0.638 (0.108) | 0.477 (0.064) | 0.731 (0.279) | 0.677

4. Secondary Outcome: Number of Participants With Change in Patient Reported Pain as Measured by Brief Pain Index
Description: The Brief Pain Index uses a scale of 0-10 to rate the severity of pain. A rating of 0 indicates no pain. A rating of 10 indicates the worst pain imaginable.
Time Frame: Cycle 1-Day 1 and Cycle 2-Day 1. Each cycle lasted 35 days.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 0.75 GBq Cohort | 1.5 GBq Cohort | 2.0 GBq Cohort | 3.0 GBq Cohort | 4.5 GBq Cohort | 6.0 GBq Cohort | 7.5 GBq Cohort | 9.0 GBq Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 0
Participants
  Change in rating of pain at its worst in the past 24 hours from Cycle 1-Day 1 to Cycle 2-Day 1: Experienced an increase in reported pain | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Change in rating of pain at its worst in the past 24 hours from Cycle 1-Day 1 to Cycle 2-Day 1: Experienced a decrease in reported pain | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Change in rating of pain at its worst in the past 24 hours from Cycle 1-Day 1 to Cycle 2-Day 1: Experienced no change in reported pain | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
  Change in rating of average pain from Cycle 1-Day 1 to Cycle 2-Day 1: Experienced an increase in reported pain | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change in rating of average pain from Cycle 1-Day 1 to Cycle 2-Day 1: Experienced a decrease in reported pain | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Change in rating of average pain from Cycle 1-Day 1 to Cycle 2-Day 1: Experienced no change in reported pain | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0

5. Secondary Outcome: Assessment of Pharmacokinetics of CTT1403
Description: The distribution half-life and the elimination half-life of CTT1403 were calculated.
Time Frame: Samples were collected during Cycle 1 (timepoints start at the initiation of infusion): Day 1 (30 min +/- 5 min and 2 hrs +/- 30 min), Day 2 (24 hrs +/- 12 hrs), Day 3 (48 hrs +/- 12 hrs), Day 8 (168 hrs +/- 24 hrs), Day 15 (336 hrs +/- 24 hrs)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 0.75 GBq Cohort | 1.5 GBq Cohort | 2.0 GBq Cohort | 3.0 GBq Cohort | 4.5 GBq Cohort | 6.0 GBq Cohort | 7.5 GBq Cohort | 9.0 GBq Cohort
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 3 | 3 | 1
hours
  Distribution half-life: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 2 | 0 | 0
  Distribution half-life |  | 0.747 | 1.044 | 0.699 (0.267) | 0.813 (0.068) | 0.680 (0.149) |  |
  Elimination half-life: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 2 | 0 | 0
  Elimination half-life |  | 28.881 | 23.902 | 29.616 (2.673) | 36.867 (4.531) | 38.173 (11.365) |  |

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected throughout the course of the study and up to 6 months after the last administered dose of the study drug, up to a total of 7 months.
Arm/Group | 0.75 GBq Cohort | 1.5 GBq Cohort | 2.0 GBq Cohort | 3.0 GBq Cohort | 4.5 GBq Cohort | 6.0 GBq Cohort | 7.5 GBq Cohort | 9.0 GBq Cohort
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 3/3 | 4/4 | 3/3 | 3/3 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/3 | 1/4 | 1/3 | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 0/1 | 2/3 | 2/4 | 2/3 | 1/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.75 GBq Cohort (N=1) | 1.5 GBq Cohort (N=1) | 2.0 GBq Cohort (N=1) | 3.0 GBq Cohort (N=3) | 4.5 GBq Cohort (N=4) | 6.0 GBq Cohort (N=3) | 7.5 GBq Cohort (N=3) | 9.0 GBq Cohort (N=1)
Grade 3 Fall (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Unrelated to study drug. Met reporting criteria per protocol due to hospitalization.
Grade 3 Syncope (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Unrelated to study drug. Met reporting criteria per protocol due to hospitalization.
Grade 3 Atrial Fibrillation with Rapid Ventricular Response (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Unrelated to study drug. Met reporting criteria per protocol due to hospitalization.
Grade 3 Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Unrelated to study drug. Met reporting criteria per protocol due to hospitalization.
Grade 3 Hyponatremia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Unrelated to study drug. Met reporting criteria per protocol due to hospitalization.
Grade 3 Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Unrelated to study drug. Met reporting criteria per protocol due to hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.75 GBq Cohort (N=1) | 1.5 GBq Cohort (N=1) | 2.0 GBq Cohort (N=1) | 3.0 GBq Cohort (N=3) | 4.5 GBq Cohort (N=4) | 6.0 GBq Cohort (N=3) | 7.5 GBq Cohort (N=3) | 9.0 GBq Cohort (N=1)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 — Number of patients that experienced Grade 1 or 2
Dry heave (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Abdominal malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Decreased apetite (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Blood in urine (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Number of patients that experienced Grade 1 or 2
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Number of patients that experienced Grade 1 or 2
Vomitting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Diaphoresis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Taste changes (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Periorbital swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Intermittent bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Number of patients that experienced Grade 1 or 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Number of patients that experienced Grade 1 or 2

LIMITATIONS AND CAVEATS:
The highest administered dose of CTT1403 was 9.0 GBq. At the 9.0 GBq dose, patients had to remain in-patient (in hospital) after administration due to continued radioactivity and for the safety of others until radioactivity dropped to an acceptable level as deemed by the hospital radiation safety committee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results for a period that is less than or equal to 45 days prior to submission for publication or disclosure to a third party. If sponsor believes patentable subject matter is disclosed, it shall, within 30 days of receipt, notify university and publication or disclosure will be withheld for a period of up to 90 days from date of receipt or until university and sponsor agree that no patentable invention exists, whichever period is shorter.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT03822871/Prot_SAP_000.pdf